CLINICAL TRIAL: NCT05391776
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TST002 Intervenous Injection in Postmenopausal Women and Men With Reduced Bone Mineral Density
Brief Title: TST002 Intervenous Injection in Postmenopausal Women and Men With Reduced Bone Mineral Density
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HJB (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TST002-1001
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A single ascending dose of TST002 Intervenous Injection (Experimental): Four single dose cohorts are designed in this study, 8 subjects will be enrolled in each cohort, Subjects in each dose group were randomized to receive TST002 or placebo in a ratio of 3:1.
  Interventions: Drug: TST002 Injection
- A single ascending dose of placebo Intervenous Injection (Placebo Comparator): Four single dose cohorts are designed in this study, 8 subjects will be enrolled in each cohort, Subjects in each dose group were randomized to receive TST002 or placebo in a ratio of 3:1.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TST002 Injection — This single dose study, ascending with phase I dose-escalation principles from 200mg up to 1200mg.
  Other Names: TST002-IgG4
  Arms: A single ascending dose of TST002 Intervenous Injection
Drug: placebo — This single dose study, ascending with phase I dose-escalation principles from 200mg up to 1200mg.
  Arms: A single ascending dose of placebo Intervenous Injection

SUMMARY:
This is a placebo-controlled, single-ascending dose, multicenter Phase I clinical study to evaluate the safety, tolerability, PK and PD characteristics of a single intravenous infusion of TST002 in subjects with reduced bone mineral density.

DETAILED DESCRIPTION:
Four single dose cohorts are designed in this study, ascending with phase I dose-escalation principles as following: 200mg, 400mg (100%), 800mg (100%), and 1200mg (50%). 8 subjects will be enrolled in each cohort, 6 for TST002 injection and 2 for placebo. Only ≤3 male subjects could be enrolled in each cohort. Subjects in each dose group were randomized to receive TST002 or placebo in a ratio of 3:1.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion and exclusion criteria to be enrolled in this study:

1. Voluntarily signe the informed consent, could walk freely, understood the study and is willing to follow it, and could complete all test procedures as planned;
2. Body mass index (BMI) : 18.0-30.0 kg/m2 (inclusive), weight ≥45 kg, BMI= weight (kg)/height 2 (m2);
3. 45-70 years old (inclusive) postmenopausal women who have been in post-menopause for 2 years or more. Menopause is defined as: 1) no spontaneous vaginal bleeding or bleeding for more than 12 months; 2) More than 1 year after bilateral oophorectomy (time for unilateral oophorectomy is calculated according to natural menopause); 3) Hysterectomy: more than 50 years old, serum FSH level & GT; 40 iu/L. 50-75 years old (inclusive) men. Male subjects should agree to use effective, investigator-approved contraceptive methods from the time they sign the informed consent until 3 months after administration.
4. BMD T score at lumbar vertebra L1-L4, total hip or femoral neck < -1.0;
5. Subjects had at least two consecutive vertebrae in L1-L4 and at least one hip bone available for dual-energy DXA bone mineral density assessment;
6. Prior to enrollment, the investigator assessed the subjects to have no medical conditions that would significantly affect the study or may increase additional health risks by asking for medical history, physical examination, and supplementary examination. If the subjects have abnormal examination reports, they can only be enrolled if the investigator evaluates that they do not pose a safety risk to the subjects or do not interfere with the safety evaluation of the clinical study, and explains the reasons.

Exclusion Criteria:

1. Blood donation or bleeding of 400mL or more within 3 months before screening; History of blood transfusion within 3 months prior to screening;
2. People who have a history of drug allergy or allergic constitution;
3. Received systemic glucocorticoid treatment 3 months before screening, and took prednisone equivalent of more than 5mg per day for a total of more than 10 days; Inhalation or topical administration within 2 weeks prior to screening is not included;
4. Have a history of alcohol or drug abuse or tobacco abuse in the past year (smoking more than 5 cigarettes per day).

   Note: Criteria for alcohol intake: weekly alcohol intake < 14 units/week, 1 unit =360 mL beer; Or 150 mL wine; Or 45 mL white wine;
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is greater than 1.25 times the upper limit of normal value or total bilirubin is greater than 1.1 times the upper limit of normal value; Renal function laboratory examination is judged to be clinically significant by researchers.
6. History of breast cancer (female subjects only); Hereditary family history of breast cancer or known BRCA1/2 gene mutation; Mammography within 6 months prior to screening does not exclude breast cancer.
7. Have a history of thrombocytopenia, or have a platelet count below the lower limit of the normal range during screening;
8. It is clinically significant to have previous diseases or hemorrhagic diseases leading to coagulation abnormalities or coagulation abnormalities during screening period;
9. Those who had a serious injury or major surgical operation within 1 month prior to the screening period, or who planned to have surgery during the study period;
10. History of solid organ and bone marrow transplants;
11. Participated in any clinical trials within 3 months prior to screening.
12. Other conditions that, in the investigator's judgment, are unsuitable for study participation, such as factors that, in the investigator's judgment, pose a risk to the safety of the subject or interfere with the study evaluation, procedure, or completion.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-04-28 (Estimated); Study Completion 2023-06-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Adverse events were collected from the time informed consent was signed until 12 weeks after the end of treatment
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

SECONDARY OUTCOMES:
Tmax | 2 hours before treatment and 12 weeks after treatment
  Time to Maximum Observed Concentration of TST002.
Cmax | 2 hours before treatment and 12 weeks after treatment.
  Maximum Observed Concentration of TST002
T1/2 | 2 hours before treatment and 12 weeks after treatment.
  Half-life Associated With the Terminal Phase of Elimination for TST002
P1NP | 2 hours before treatment and days 8,29,43,57 and 85
  Percent Change From Baseline in Procollagen TYpe 1 N-terminal Propeptide
BDM | baseline and day 85
  Percent change from baseline in Bone Mineral Density at L1-L4,total hip and femoral neck
Immunogenicity | 2 hours before treatment and days 15,29 and 85
  Positive rate and timing of anti-TST002 antibody and neutralizing antibody
Serum total osteostatin | 2 hours before treatment and 12 weeks after treatment
  Percent change from baseline in serum total sclerostin
CL | 2 hours before treatment and 12 weeks after treatment
  System clearance rate of TST002

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - West China Hospital，Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No